CLINICAL TRIAL: NCT01337713
Title: Efficacy of Massage and Light Touch Therapy for the Treatment of Generalized Anxiety Disorder
Brief Title: Efficacy of Massage Therapy in the Treatment of Generalized Anxiety Disorder (GAD)
Acronym: GAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mark H. Rapaport, Professor and Chair, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00052054; 7R21AT004208-02 (NIH)
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Generalized Anxiety Disorder
Keywords: Anxiety, GAD, Massage
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Swedish Massage (Experimental)
  Interventions: Other: Swedish Massage
- Light Touch (Sham Comparator)
  Interventions: Other: Light Touch

INTERVENTIONS:
Other: Swedish Massage — Swedish massage, 45 minutes, 2 x per week for 6 weeks
  Arms: Swedish Massage
Other: Light Touch — Light touch, 45 minutes, 2 x week for 6 weeks
  Arms: Light Touch

SUMMARY:
There is an impressive and growing body of data suggesting that massage therapy is effective in decreasing some symptoms of pathological conditions as well as facilitating growth, reducing pain, increasing alertness, diminishing symptoms of depression and anxiety, and enhancing immune function. Preliminary studies suggest that massage therapy decreases symptoms of anxiety and depression, and lowers salivary cortisol levels in a wide array of childhood and adult neuropsychiatric disorders including post-traumatic stress disorder, attention-deficit-disorder hyperactivity, depression, bulimia and anorexia-nervosa. Generalized Anxiety Disorder (GAD) is characterized by the presence of a constellation of signs and symptoms for at least 6 months in duration, with some type of functional disability or decrease in quality of life. The signs and symptoms of GAD include a myriad of somatic symptoms including muscle tension, headaches, backaches, fatigue, restlessness, insomnia, as well as psychological feelings of worry, anxiety, and feeling overwhelmed. Both pharmacotherapy and psychotherapy are effective in decreasing the signs and symptoms of GAD. Unfortunately, the vast majority of patients with GAD never receive adequate pharmacotherapy or psychotherapy. Therefore, the development of a complementary and alternative therapy that has demonstrated efficacy for GAD might be well received by patients.

This study's goals are to investigate the efficacy of Swedish massage therapy vs. light touch therapy and better understand the biological effects of massage in patients with anxiety. Qualified participants will be randomly assigned to one of two groups in which they will receive Swedish massage therapy twice per week for 12 weeks or Light Touch therapy twice per week for 6 weeks followed by Swedish massage therapy twice per week for the next 6 weeks. The total length of the study is 13 weeks, which includes a screening visit that takes about 3 hours and two therapy visits per week for 12 weeks that last about 1 hour each. Blood and urine will be collected at three of the visits. Compensation is up to $400 for completing the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old
* Able to read and understand English
* Medically healthy as demonstrated by a normal history and physical examination
* Meet criteria for a primary diagnosis of current GAD as demonstrated by a structured clinical interview for DSM-IV (SCID),
* HAM-A score of greater than 14
* Normal blood work and urinalysis (CBC, Renal, Hepatic, Tox Screen)

Exclusion Criteria:

* Individuals who lack a capacity to consent, or whose capacity to provide consent is questionable to the investigator
* Current suicidal ideation (core of 3 or more on the HAM-D suicide item)
* Current diagnosis of schizophrenia
* Current diagnosis of bipolar disorder
* Current diagnosis of borderline personality disorder
* Comorbid secondary disorder diagnosis of OCD
* Current illicit drug use
* Excessive regular use of alcohol (more than two 5-oz glasses of wine or equivalents/day) or a history of binge drinking (more than 7 drinks/24 hour period) within the last six months
* Regular or "PRN" psychotropic medication use
* Current participation in psychotherapy or cognitive behavioral therapy
* Pregnancy
* Shift work schedule
* Active dieting for weight loss
* Active medical problems
* Fibromyalgia (on daily medication)
* Arthritis requiring daily meds and unable to abstain from meds for duration of study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale | 25 times over an average of 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Rapaport, M.D., Principal Investigator — Emory University
Locations (1):
- Emory University, Department of Psychiatry, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Rapaport MH, Schettler P, Larson ER, Edwards SA, Dunlop BW, Rakofsky JJ, Kinkead B. Acute Swedish Massage Monotherapy Successfully Remediates Symptoms of Generalized Anxiety Disorder: A Proof-of-Concept, Randomized Controlled Study. J Clin Psychiatry. 2016 Jul;77(7):e883-91. doi: 10.4088/JCP.15m10151. PMID 27464321